CLINICAL TRIAL: NCT01971697
Title: Short Term Socio-economic Impact Due to Blunt Orthopedics Trauma on the Victims in Uganda
Brief Title: Socio-Economic Survey in Uganda
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00046624
Record Dates: First submitted 2013-07-15; First posted 2013-10-29 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-05

CONDITIONS: Orthopaedic Injury

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will be conducted at Mulago Teaching Hospital. Patients coming to the ER with an orthopaedic injury will be approached. If a patient consents to be part of the study, they will complete a questionnaire. Participation in the study will end as soon as the questionnaire is completed.

DETAILED DESCRIPTION:
All patients will be recruited from the orthopedics inpatient wards and emergency department at Mulago National Referral Hospital. Only patients who have sustained an orthopedics injury will be included in this study, and the severity will be recorded for future references. No Protected Health Information (PHI) will be collected throughout the study.

Steps

1. Identify patients from Mulago Teaching Hospital
2. Enrollment of patients into survey study
3. Administer survey to patients at 1st meet up
4. Administer survey to doctor-in-charge?
5. Compilations of survey results into excel spreadsheet. Participants will be assigned an ID. The study team does not intend to collect any PHI.
6. Statistical Analysis.

ELIGIBILITY:
Inclusion criteria:

* Subject is a male or female 18 years old or older.
* all patients presented at Mulago National Referral Hospital with orthopedics trauma injuries regardless of age and gender.

Exclusion criteria:

- patients presented with all other conditions other than orthopedics related injuries that may require long term care. Some examples are head injuries leading to long term damage, loss of sights, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Urgent care patients. Patients coming to the ER with a orthopaedic injury.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Immediate social-economic impact of orthopedics trauma as measured by socio-Economic Questionnaire | approximately 20 minutes
  A short socio-economic questionnaire will be provided to all enrolled patients

CONTACTS AND LOCATIONS:
Overall Officials: William Richadson, MD, Principal Investigator — Duke University
Locations (2):
- Duke University Medical Center, Durham, North Carolina, United States
- Mulago National Referral Hospital, Kampala, Uganda